CLINICAL TRIAL: NCT01536470
Title: Effectiveness of Noradrenaline to Control Intraoperative Arterial Pressure in High-risk Surgical Patients: A Multicentre Prospective Randomized Controlled Trial
Brief Title: Intraoperative Noradrenaline to Control Arterial Pressure (INPRESS Study)
Acronym: INPRESS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Aguettant laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHU-0111; 2011-004232-66 (EudraCT Number)
Record Dates: First submitted 2012-02-13; First posted 2012-02-22 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Control of Arterial Blood Pressure
Keywords: Intraoperative hemodynamic; Arterial pressure; Postoperative complications; Intraoperative fluids; Noradrenaline
MeSH Terms: conditions — Postoperative Complications | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noradrenaline (Experimental): Continuous infusion of noradrenaline to maintain arterial blood pressure management in high-risk surgical patients
  Interventions: Other: noradrenaline
- Ephedrine chorhydrate (Experimental): Conventional treatment of hypotension (defined as a blood pressure of below 80 mmHg or a decrease of more than 40% from baseline)using intravenous bolus of Ephedrine chorhydrate
  Interventions: Other: Ephedryne chorydrate

INTERVENTIONS:
Other: noradrenaline — The primary objective of the study is to compare two strategies of intraoperative blood pressure management in high-risk surgical patients: 1- Continuous infusion of noradrenaline to maintain arterial blood pressure of no more than 10% below its baseline value; 2- Conventional treatment of hypotension (defined as a blood pressure of below 80 mmHg or a decrease of more than 40% from baseline) using intravenous bolus of Ephedrine chorhydrate.
  Arms: Noradrenaline
Other: Ephedryne chorydrate
  Arms: Ephedrine chorhydrate

SUMMARY:
The purpose of this study is to evaluate whether a preventive strategy of intraoperative arterial hypotension using noradrenaline can reduce the incidence of postoperative organ failure.

DETAILED DESCRIPTION:
The maintenance of arterial blood pressure is essential for organ perfusion pressure. Intraoperative hypotension is a frequent complication both after induction and during maintenance of anaesthesia, ranging from 5% to 75% depending on the chosen definition. Tissue hypoperfusion exposes to the occurrence of a systemic inflammatory response syndrome and is a key determinant of postoperative complications. Persistent intraoperative hypotension has been reported as an important prognostic factor of postoperative morbidity and mortality. Adequate treatment of arterial hypotension is therefore of particular importance during surgery, but optimal strategy of intraoperative blood pressure management remains undetermined, especially in high-risk patients. Target ranges for arterial pressure are not clearly defined, and hypotension is usually defined as a systolic pressure of less than 80 mmHg or a decrease of more than 40% from baseline.

Traditionally, management of intraoperative hypotension consisted primarily of fluid administration whereas vasoconstrictors, such as Ephedrine chlorhydrate, are often used as a second line therapy. This may, however, expose patients to prolonged hypotension and to excessive fluid administration, and each of them may alter tissue oxygenation.

Recent experimental data have shown that noradrenaline, which has - and -adrenergic effects, has no detrimental effects on microcirculatory blood flow and tissue oxygenation in the intestinal tract. Because of anaesthesia-induced vasodilatation, the use of a continuous infusion of noradrenaline to increase systemic vascular resistance could be useful to prevent detrimental effects of compromised tissue perfusion, especially in high-risk surgical patients.

The primary objective of the study is to compare two strategies of intraoperative blood pressure management in high-risk surgical patients: 1- Continuous infusion of noradrenaline to maintain arterial blood pressure of no more than 10% below its baseline value; 2- Conventional treatment of hypotension (defined as a blood pressure of below 80 mmHg or a decrease of more than 40% from baseline) using intravenous bolus of Ephedrine chorhydrate.

The investigators hypothesis is that maintenance of arterial blood pressure with noradrenaline could reduce postoperative organ dysfunction in high-risk surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* ASA score ≥ 2
* Planned and unplanned surgical procedures
* Abdominal, orthopaedic and vascular surgery
* Expected duration ≥ 2 hours
* AKI risk index ≥ class 3

Exclusion Criteria:

* Severe preoperative hypertension (not controlled)
* Creatinine clearance < 30 ml/min or preoperative dialysis
* Acute cardiac failure
* Preoperative sepsis
* Preoperative hemodynamic failure (shock)
* Intraoperative use of locoregional anaesthesia (epidural and spinal)
* Patient refusal
* Pregnancy and/or lactation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of postoperative SIRS and at least one major organ dysfunction | day-7

SECONDARY OUTCOMES:
Incidence of intraoperative hypotension | at day 7
Incidence of intraoperative hypertension | at day 7
Incidence of intraoperative bradycardia | at day 7
Intraoperative volume of fluid perfused | at day 7
Intraoperative blood losses | at day 7
Need for intraoperative transfusion | at day 7
Postoperative organ failure | at day 7
Biologic criteria: plasma concentration of NGAL, creatinine, CRP, serum lactate, troponine) | at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel FUTIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Futier E, Lefrant JY, Guinot PG, Godet T, Lorne E, Cuvillon P, Bertran S, Leone M, Pastene B, Piriou V, Molliex S, Albanese J, Julia JM, Tavernier B, Imhoff E, Bazin JE, Constantin JM, Pereira B, Jaber S; INPRESS Study Group. Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357. doi: 10.1001/jama.2017.14172. PMID 28973220